CLINICAL TRIAL: NCT05838612
Title: Short-term Warm Water Immersion as a Heat Acclimation Strategy to Enhance Heat Dissipation in Older Adults: An Exploratory Study
Brief Title: Hot Water Immersion as a Heat Acclimation Strategy in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, Principal Investigator, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HEPRU-2023-02
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Hyperthermia; Heat Exposure; Heat Stress; Thermoregulation; Aging
Keywords: Thermoregulation; Warm-water immersion; Heat acclimation; Aging
MeSH Terms: conditions — Hyperthermia; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Each participant will complete seven consecutive experimental sessions consisting of a passive heat acclimation involving a one hour immersion in warm water (~40°C) with core temperature clamped at 38.5°C. Prior to and following the passive heat acclimation protocol, study participants will perform an exercise-heat stress test (Days 0 and 8) to assess whole-body heat loss in a hot-dry environment (40°C, 15% relative humidity). The exercise protocol will consist of three successive 30-minute bouts of exercise performed at increasing rates of metabolic heat production (i.e., 150, 200 and 250 W/m2), each separated by a 15-minute rest break, with the final recovery 1-hour in duration.
Masking Description: Data will be blinded prior to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat Acclimation (Experimental): Participants will undergo an exercise heat stress test prior to and following seven consecutive days of warm-water immersion (~40°C) of 1-hour duration with core temperature clamped at 38.5°C. During the exercise-heat stress test participants will perform three, successive 30-minute bouts of semi-recumbent cycling performed at increasing fixed loads of metabolic heat production of 150, 200 and 250 W/m2 (i.e., exercise bout 1, exercise bout 2 and exercise bout 3, respectively), each separated by 15-minute of rest break with the final recovery extended to 1-hour.
  Interventions: Other: Heat acclimation

INTERVENTIONS:
Other: Heat acclimation — Participants will complete a 7-day passive heat acclimation protocol consisting of immersion in warm water (~40°C) for 1 hour over 7 consecutive days.

SUMMARY:
Aging is associated with impairments in heat loss responses of skin blood flow and sweating leading to reductions in whole-body heat loss. Consequently, older adults store more body heat and experience greater elevations in core temperature during heat exposure at rest and during exercise. This maladaptive response occurs in adults as young as 40 years of age. Recently, heat acclimation associated with repeated bouts of exercise in the heat performed over 7 successive days has been shown to enhance whole-body heat loss in older adults, leading to a reduction in body heat storage. However, performing exercise in the heat may not be well tolerated or feasible for many older adults. Passive heat acclimation, such as the use of warm-water immersion may be an effective, alternative method to enhance heat-loss capacity in older adults. Thus, the following study aims to assess the effectiveness of a 7-day warm-water immersion (~40°C) protocol in enhancing whole-body heat loss in older adults. Warm-water immersion will consist of a one-hour immersion in warm water with core temperature clamped at 38.5°C. Improvements in whole-body heat loss will be assessed during an incremental exercise protocol performed in dry heat (i.e., 40°C, ~15% relative humidity) prior to and following the 7-day passive heat acclimation protocol. The incremental exercise protocol will consist of three 30 minute exercise bouts performed at increasing fixed rates of metabolic heat production (i.e., 150, 200, and 250 W/m2), each separated by 15-minutes of recovery, with exception final recovery will be 1-hour in duration) performed in a direct calorimeter (a device that provides a precise measurement of the heat dissipated by the human body).

ELIGIBILITY:
Inclusion Criteria:

* Elderly (60-80 years), non-smoking adults.
* Not engaged in regular physical activity (>2 sessions/week for ≥20 minutes per session).
* Willing to provide informed consent.
* Healthy, no diagnosed health conditions.
* Body Mass index (BMI) <35 kg/m2.

Exclusion Criteria:

* Heat adapted due to repeated exposure to hot environments within the last 3 weeks (use sauna, recent travel to hot climates, other).

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Evaporative heat loss | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Evaporative heat loss as assessed using a direct air calorimeter.
Evaporative heat loss | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Evaporative heat loss as assessed using a direct air calorimeter.
Evaporative heat loss | End of 30 minute bout 3 (average of last 5 minutes).
  Evaporative heat loss as assessed using a direct air calorimeter.
Whole-body heat loss | End of 30 minute exercise bout 1 (average of last 5 minutes).
  The sum of evaporative and dry heat exchange will be quantified during each exercise period (i.e., 150, 200 and 250 W/m2).
Whole-body heat loss | End of 30 minute exercise bout 2 (average of last 5 minutes).
  The sum of evaporative and dry heat exchange will be quantified during each exercise period (i.e., 150, 200 and 250 W/m2).
Whole-body heat loss | End of 30 minute exercise bout 3 (average of last 5 minutes).
  The sum of evaporative and dry heat exchange will be quantified during each exercise period (i.e., 150, 200 and 250 W/m2).

SECONDARY OUTCOMES:
Body heat storage | Change from start to end of 30 minute exercise bout 1
  Cumulative amount of heat stored within the body calculated as the temporal summation of metabolic heat production and net heat loss.
Body heat content | Change from start to end of 30 minute exercise bout 2
  Cumulative amount of heat stored within the body calculated as the temporal summation of metabolic heat production and net heat loss.
Body heat storage | Change from start to end of 30 minute exercise bout 3
  Cumulative amount of heat stored within the body calculated as the temporal summation of metabolic heat production and net heat loss.
Cumulative body heat storage | Change from baseline resting to end of exercise bout 3
  Cumulative amount of heat stored within the body calculated as the temporal summation of metabolic heat production and net heat loss.
Dry heat loss | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Dry heat loss as assessed using a direct air calorimeter.
Dry heat loss | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Dry heat loss as assessed using a direct air calorimeter.
Dry heat loss | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Dry heat loss as assessed using a direct air calorimeter.
Core temperature | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Core temperature indexed by rectal/visceral temperature
Core temperature | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Core temperature indexed by rectal/visceral temperature
Core temperature | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Core temperature indexed by rectal/visceral temperature
Change in core temperature | Change from baseline resting to end of end of 30 minute exercise bout 3.
  Core temperature indexed by rectal/visceral temperature
Skin temperature | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Skin temperature measured at 4-sites (chest, upper arm, thigh, calf) with mean value calculated as weighted value of 4 sites - upper arm, 30%; chest, 30%; thigh, 20%; and calf, 20%.
Skin temperature | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Skin temperature measured at 4-sites (chest, upper arm, thigh, calf) with mean value calculated as weighted value of 4 sites - upper arm, 30%; chest, 30%; thigh, 20%; and calf, 20%.
Skin temperature | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Skin temperature measured at 4-sites (chest, upper arm, thigh, calf) with mean value calculated as weighted value of 4 sites - upper arm, 30%; chest, 30%; thigh, 20%; and calf, 20%.
Change in skin temperature | Change from baseline resting to end of end of 30 minute exercise bout 3.
  Skin temperature measured at 4-sites (chest, upper arm, thigh, calf) with mean value calculated as weighted value of 4 sites - upper arm, 30%; chest, 30%; thigh, 20%; and calf, 20%.
Heart rate | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Measured continuously with chest-band device
Heart rate | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Measured continuously with chest-band device
Heart rate | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Measured continuously with chest-band device
Heart rate variability | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Measures of variability computed from the time, frequency, time-frequency, scale-invariant, entropy, and other nonlinear domains
Heart rate variability | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Measures of variability computed from the time, frequency, time-frequency, scale-invariant, entropy, and other nonlinear domains
Heart rate variability | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Measures of variability computed from the time, frequency, time-frequency, scale-invariant, entropy, and other nonlinear domains
Thermal comfort scale | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Thermal comfort assessed via a questionnaire using the ASHRAE 4-point scale ("1=comfortable to 4=very uncomfortable")
Thermal comfort scale | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Thermal comfort assessed via a questionnaire using the ASHRAE 4-point scale ("1=comfortable to 4=very uncomfortable")
Thermal comfort scale | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Thermal comfort assessed via a questionnaire using the ASHRAE 4-point scale ("1=comfortable to 4=very uncomfortable")
Thermal sensation scale | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Thermal sensation will be assessed using the ASHRAE 7-point scale ("0=neutral to 7=extremely hot")
Thermal sensation scale | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Thermal sensation will be assessed using the ASHRAE 7-point scale ("0=neutral to 7=extremely hot")
Thermal sensation scale | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Thermal sensation will be assessed using the ASHRAE 7-point scale ("0=neutral to 7=extremely hot")
Thirst sensation scale | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Thirst sensation will be quantified using a 9-point scale ("1=not thirsty at all to 9=very, very thirsty")
Thirst sensation scale | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Thirst sensation will be quantified using a 9-point scale ("1=not thirsty at all to 9=very, very thirsty")
Thirst sensation scale | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Thirst sensation will be quantified using a 9-point scale ("1=not thirsty at all to 9=very, very thirsty")
Rating of perceived exertion | End of 30 minute exercise bout 1 (average of last 5 minutes).
  Rating of perceived exertion will be quantified using a 14-point scale ("6=no exertion at all to 20=maximal exertion")
Rating of perceived exertion | End of 30 minute exercise bout 2 (average of last 5 minutes).
  Rating of perceived exertion will be quantified using a 14-point scale ("6=no exertion at all to 20=maximal exertion")
Rating of perceived exertion | End of 30 minute exercise bout 3 (average of last 5 minutes).
  Rating of perceived exertion will be quantified using a 14-point scale ("6=no exertion at all to 20=maximal exertion")

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD., Principal Investigator — University of Ottawa
Locations (1):
- Univerisity of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available with approved analysis plan and signed access agreement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following publication of the main study report(s)
Access Criteria: Approved analysis plan and signed access agreement

REFERENCES:
- [Derived] Janetos KT, O'Connor F, Morris N, Kenny GP. The influence of heat acclimation on the relation and agreement between perceptual and physiological strain in older males during exercise-heat stress. Appl Physiol Nutr Metab. 2026 Jan 16. doi: 10.1139/apnm-2025-0360. Online ahead of print. PMID 41549363
- [Derived] Janetos KT, O'Connor FK, Meade RD, Richards BJ, Koetje NJ, Kirby NV, McCormick JJ, Flouris AD, Kenny GP. Short-Term Warm Water Immersion for Improving Whole-Body Heat Loss in Older Men. Med Sci Sports Exerc. 2025 Jun 1;57(6):1137-1147. doi: 10.1249/MSS.0000000000003649. Epub 2025 Jan 17. PMID 39820413